CLINICAL TRIAL: NCT02898129
Title: Evaluating the Relationship Between Environmental Risk Factors in Housing Types and Chronic Respiratory Diseases in Ho Chi Minh City
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brugmann University Hospital (Other)
Responsible Party: Principal Investigator, Olivier Michel, Head of clinic, Brugmann University Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: CHUB-CRD-Housing
Record Dates: First submitted 2016-09-08; First posted 2016-09-13 (Estimated); Last update posted 2017-08-04 (Actual); Status verified 2017-08

CONDITIONS: Chronic Respiratory Diseases
Keywords: chronic respiratory diseases; housing; lung function test
MeSH Terms: interventions — Surveys and Questionnaires; Respiratory Function Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Tube houses (Experimental): Tube Houses. Group of 75-100 houses, with 4 inhabitants per house. Expected number of participants: 300-400. Predicted number of non-smoker chronic respiratory disease of 18-24.
  Interventions: Other: Questionnaire; Device: Lung function test
- Apartment (Experimental): Apartments. Group of 75-100 apartments, with 4 inhabitants per apartment. Expected number of participants: 300-400. Predicted number of non-smoker chronic respiratory disease of 18-24.
  Interventions: Other: Questionnaire; Device: Lung function test
- Rental Houses (Experimental): Rental Houses. Group of 150-200 rental houses, with 2 inhabitants per rental house. Expected number of participants: 300-400. Predicted number of non-smoker chronic respiratory disease of 18-24.
  Interventions: Other: Questionnaire; Device: Lung function test
- Rural houses (Experimental): Rural Houses. Group of 40-60 rural houses, with 5 inhabitant per rural house. Expected number of participants: 200-300. Predicted number of non-smoker chronic respiratory disease of 12-18.
  Interventions: Other: Questionnaire; Device: Lung function test

INTERVENTIONS:
Other: Questionnaire
Device: Lung function test — Basic lung function test performed with a micro-spirometer, without broncho dilatator

SUMMARY:
The research question is "Are the different types of house in Ho Chi Minh city equally contributing to chronic respiratory diseases?".

According to this question, a cross-sectional and explorative study was set up to explore the differences in the environmental characteristics and prevalence of chronic respiratory diseases among common housing types in Ho Chi Minh city. Preliminary work was performed in 100 houses (20 houses per type, included tube houses, rental houses, rural houses, slum and apartment) from November 2013 to June 2015. It included measures by environmental devices, questionnaires and indoor activities diaries.

This study will aim to collect information about the prevalence of chronic respiratory diseases (CRDs) inside those house types to understand more about role of house types in developing CRDs.

The objective is:

1. to evaluate the relationships between the type of house and lung function of inhabitants in each housing type.
2. to evaluate the effects of environmental risk factors in each house type on prevalence of CRDs

ELIGIBILITY:
Inclusion Criteria:

* Everybody

Exclusion Criteria:

* Not able to answer the questionnaire or give informed consent
* Have a contra-indication for lung function test (acute myocardial infarction less that 1 month ago, pain related to spirometry, dementia/confused)

Ages: 10 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1500 (Actual)
Dates: Start 2016-09; Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
FEV1/FVC | 5 minutes
  Basic lung function test, without broncho dilatation (micro-spirometer). All lung function related outcomes are performed during the same test. FEV1: forced expiratory volume in one second. FVC: Forced vital capacity.
FVC | 5 minutes
  Basic lung function test, without broncho dilatation (micro-spirometer). All lung function related outcomes are performed during the same test.FVC: Forced vital capacity.
VC | 5 minutes
  Basic lung function test, without broncho dilatation (micro-spirometer). All lung function related outcomes performed during the same test. VC: Vital capacity
FEF 25-75% | 5 minutes
  Basic lung function test, without broncho dilatation (micro-spirometer).All lung function related outcomes are performed during the same test. FEF: Forced expiratory flow
Socio-demographic status | around 10 minutes
  Socio-demographic data, assessed by a home made questionnaire
Health status | around 10 minutes
  Health status (symptomatology) data, assessed by a home made questionnaire
Indoor air exposure time | around 10 minutes
  Indoor air exposure (time spent indoor within housing types, with associated air characteristics) data, assessed by a home made questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Pham Ngoc Thach University of medicine, Ho Chi Minh City, Vietnam

REFERENCES:
- [Background] Pellegrino R, Viegi G, Brusasco V, Crapo RO, Burgos F, Casaburi R, Coates A, van der Grinten CP, Gustafsson P, Hankinson J, Jensen R, Johnson DC, MacIntyre N, McKay R, Miller MR, Navajas D, Pedersen OF, Wanger J. Interpretative strategies for lung function tests. Eur Respir J. 2005 Nov;26(5):948-68. doi: 10.1183/09031936.05.00035205. No abstract available. PMID 16264058
- [Background] Lung function testing: selection of reference values and interpretative strategies. American Thoracic Society. Am Rev Respir Dis. 1991 Nov;144(5):1202-18. doi: 10.1164/ajrccm/144.5.1202. No abstract available. PMID 1952453
- [Background] Quanjer PH, Tammeling GJ, Cotes JE, Pedersen OF, Peslin R, Yernault JC. Lung volumes and forced ventilatory flows. Report Working Party Standardization of Lung Function Tests, European Community for Steel and Coal. Official Statement of the European Respiratory Society. Eur Respir J Suppl. 1993 Mar;16:5-40. No abstract available. PMID 8499054
- [Background] Stocks J, Quanjer PH. Reference values for residual volume, functional residual capacity and total lung capacity. ATS Workshop on Lung Volume Measurements. Official Statement of The European Respiratory Society. Eur Respir J. 1995 Mar;8(3):492-506. doi: 10.1183/09031936.95.08030492. No abstract available. PMID 7789503
- [Background] American Thoracic Society. Single-breath carbon monoxide diffusing capacity (transfer factor). Recommendations for a standard technique--1995 update. Am J Respir Crit Care Med. 1995 Dec;152(6 Pt 1):2185-98. doi: 10.1164/ajrccm.152.6.8520796. No abstract available.
- [Background] Cotes JE, Chinn DJ, Quanjer PH, Roca J, Yernault JC. Standardization of the measurement of transfer factor (diffusing capacity). Report Working Party Standardization of Lung Function Tests, European Community for Steel and Coal. Official Statement of the European Respiratory Society. Eur Respir J Suppl. 1993 Mar;16:41-52. No abstract available. PMID 8499053
- [Background] Wang X, Dockery DW, Wypij D, Fay ME, Ferris BG Jr. Pulmonary function between 6 and 18 years of age. Pediatr Pulmonol. 1993 Feb;15(2):75-88. doi: 10.1002/ppul.1950150204. PMID 8474788
- [Background] Quanjer PH, Stocks J, Polgar G, Wise M, Karlberg J, Borsboom G. Compilation of reference values for lung function measurements in children. Eur Respir J Suppl. 1989 Mar;4:184S-261S. No abstract available. PMID 2659037
- [Background] COPD-more than just tobacco smoke. Lancet. 2009 Aug 29;374(9691):663. doi: 10.1016/S0140-6736(09)61535-X. No abstract available. PMID 19716941
- [Background] Bousquet J, Kiley J, Bateman ED, Viegi G, Cruz AA, Khaltaev N, Ait Khaled N, Baena-Cagnani CE, Barreto ML, Billo N, Canonica GW, Carlsen KH, Chavannes N, Chuchalin A, Drazen J, Fabbri LM, Gerbase MW, Humbert M, Joos G, Masjedi MR, Makino S, Rabe K, To T, Zhi L. Prioritised research agenda for prevention and control of chronic respiratory diseases. Eur Respir J. 2010 Nov;36(5):995-1001. doi: 10.1183/09031936.00012610. Epub 2010 Mar 11. PMID 20223919
- [Background] Samet JM, Spengler JD. Indoor environments and health: moving into the 21st century. Am J Public Health. 2003 Sep;93(9):1489-93. doi: 10.2105/ajph.93.9.1489. PMID 12948968
- [Background] Bardana EJ Jr. Indoor pollution and its impact on respiratory health. Ann Allergy Asthma Immunol. 2001 Dec;87(6 Suppl 3):33-40. doi: 10.1016/s1081-1206(10)62338-1. PMID 11770681
- [Background] Bruce N, Perez-Padilla R, Albalak R. Indoor air pollution in developing countries: a major environmental and public health challenge. Bull World Health Organ. 2000;78(9):1078-92. PMID 11019457
- [Background] Ezzati M, Kammen DM. The health impacts of exposure to indoor air pollution from solid fuels in developing countries: knowledge, gaps, and data needs. Environ Health Perspect. 2002 Nov;110(11):1057-68. doi: 10.1289/ehp.021101057. PMID 12417475
- [Background] Smith KR. Indoor air pollution in developing countries: recommendations for research. Indoor Air. 2002 Sep;12(3):198-207. doi: 10.1034/j.1600-0668.2002.01137.x. PMID 12244750
- [Background] Smith KR, Mehta S. The burden of disease from indoor air pollution in developing countries: comparison of estimates. Int J Hyg Environ Health. 2003 Aug;206(4-5):279-89. doi: 10.1078/1438-4639-00224. PMID 12971683
- [Background] Smith KR, Samet JM, Romieu I, Bruce N. Indoor air pollution in developing countries and acute lower respiratory infections in children. Thorax. 2000 Jun;55(6):518-32. doi: 10.1136/thorax.55.6.518. PMID 10817802
- [Background] Rojas-Bracho L, Suh HH, Koutrakis P. Relationships among personal, indoor, and outdoor fine and coarse particle concentrations for individuals with COPD. J Expo Anal Environ Epidemiol. 2000 May-Jun;10(3):294-306. doi: 10.1038/sj.jea.7500092. PMID 10910121
- [Background] Sarnat JA, Koutrakis P, Suh HH. Assessing the relationship between personal particulate and gaseous exposures of senior citizens living in Baltimore, MD. J Air Waste Manag Assoc. 2000 Jul;50(7):1184-98. doi: 10.1080/10473289.2000.10464165. PMID 10939211
- [Background] Jaakkola MS. Environmental tobacco smoke and health in the elderly. Eur Respir J. 2002 Jan;19(1):172-81. doi: 10.1183/09031936.02.00270702. PMID 11852892
- [Background] Smith KR. National burden of disease in India from indoor air pollution. Proc Natl Acad Sci U S A. 2000 Nov 21;97(24):13286-93. doi: 10.1073/pnas.97.24.13286. PMID 11087870
- [Background] Briggs D. Environmental pollution and the global burden of disease. Br Med Bull. 2003;68:1-24. doi: 10.1093/bmb/ldg019. PMID 14757707
- [Background] Raw GJ, Coward SK, Brown VM, Crump DR. Exposure to air pollutants in English homes. J Expo Anal Environ Epidemiol. 2004;14 Suppl 1:S85-94. doi: 10.1038/sj.jea.7500363. PMID 15118750
- [Background] Viegi G, Simoni M, Scognamiglio A, Baldacci S, Pistelli F, Carrozzi L, Annesi-Maesano I. Indoor air pollution and airway disease. Int J Tuberc Lung Dis. 2004 Dec;8(12):1401-15. PMID 15636485
- [Background] Levesqu B, Allaire S, Gauvin D, Koutrakis P, Gingras S, Rhainds M, Prud'Homme H, Duchesne JF. Wood-burning appliances and indoor air quality. Sci Total Environ. 2001 Dec 17;281(1-3):47-62. doi: 10.1016/s0048-9697(01)00834-8. PMID 11778959
- [Background] Naeher LP, Smith KR, Leaderer BP, Neufeld L, Mage DT. Carbon monoxide as a tracer for assessing exposures to particulate matter in wood and gas cookstove households of highland Guatemala. Environ Sci Technol. 2001 Feb 1;35(3):575-81. doi: 10.1021/es991225g. PMID 11351731
- [Background] Rollin HB, Mathee A, Bruce N, Levin J, von Schirnding YE. Comparison of indoor air quality in electrified and un-electrified dwellings in rural South African villages. Indoor Air. 2004 Jun;14(3):208-16. doi: 10.1111/j.1600-0668.2004.00238.x. PMID 15104789
- [Background] Schwela D. Cooking smoke: a silent killer. People Planet. 1997;6(3):24-5. PMID 12321046
- [Background] Wolkoff P, Schneider T, Kildeso J, Degerth R, Jaroszewski M, Schunk H. Risk in cleaning: chemical and physical exposure. Sci Total Environ. 1998 Apr 23;215(1-2):135-56. doi: 10.1016/s0048-9697(98)00110-7. PMID 9599458
- [Background] Delfino RJ. Epidemiologic evidence for asthma and exposure to air toxics: linkages between occupational, indoor, and community air pollution research. Environ Health Perspect. 2002 Aug;110 Suppl 4(Suppl 4):573-89. doi: 10.1289/ehp.02110s4573. PMID 12194890
- [Background] Payne-Sturges DC, Burke TA, Breysse P, Diener-West M, Buckley TJ. Personal exposure meets risk assessment: a comparison of measured and modeled exposures and risks in an urban community. Environ Health Perspect. 2004 Apr;112(5):589-98. doi: 10.1289/ehp.6496. PMID 15064166
- [Background] Flohr C, Tuyen LN, Quinnell RJ, Lewis S, Minh TT, Campbell J, Simmons C, Telford G, Brown A, Hien TT, Farrar J, Williams H, Pritchard DI, Britton J. Reduced helminth burden increases allergen skin sensitization but not clinical allergy: a randomized, double-blind, placebo-controlled trial in Vietnam. Clin Exp Allergy. 2010 Jan;40(1):131-42. doi: 10.1111/j.1365-2222.2009.03346.x. Epub 2009 Sep 15. PMID 19758373
- [Background] Regional COPD Working Group. COPD prevalence in 12 Asia-Pacific countries and regions: projections based on the COPD prevalence estimation model. Respirology. 2003 Jun;8(2):192-8. doi: 10.1046/j.1440-1843.2003.00460.x. PMID 12753535
- [Background] Dherani M, Pope D, Mascarenhas M, Smith KR, Weber M, Bruce N. Indoor air pollution from unprocessed solid fuel use and pneumonia risk in children aged under five years: a systematic review and meta-analysis. Bull World Health Organ. 2008 May;86(5):390-398C. doi: 10.2471/blt.07.044529. PMID 18545742
- [Background] Tan WC, Ng TP. COPD in Asia: where East meets West. Chest. 2008 Feb;133(2):517-27. doi: 10.1378/chest.07-1131. PMID 18252918